CLINICAL TRIAL: NCT02532439
Title: Bone Microarchitectural Database Constitution From High Resolution Peripheral Quantitative Computed Tomography (HR-pQCT) Device in Clinical Situation Potentially Associated With Bone Loss
Brief Title: Bone Microarchitectural Database Constitution From HR-pQCT Device in Clinical Situation Potentially Associated With Bone Loss
Acronym: DMPOs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1408063; 2014-A00771-46 (Other: ANSM)
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Osteoporosis; Bone Loss
Keywords: fracture osteoporosis; bone microarchitecture; Inflammatory joint diseases; Bone fragility; Rheumatoid Arthritis; Spondyloarthritis; Primary Hyperparathyroidism; constitutional thinness; anorexia nervosa
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Osteoporotic Fractures; Arthritis, Rheumatoid; Spondylarthritis; Hyperparathyroidism, Primary; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): Measure bone quality and quantity with HR-pQCT, pQCT and DEXA of patient group Patient group is patient with one of the following pathology : Osteoporosis, Bone Fragility, articular inflammatory disease or Endocrine diseases
  Interventions: Device: HR-pQCT; Device: DEXA; Device: pQCT
- control group (Experimental): Measure bone quality and quantity with HR-pQCT, pQCT and DEXA of control group. Patient group is patient with episode of acute back pain or radicular pain
  Interventions: Device: HR-pQCT; Device: DEXA; Device: pQCT

INTERVENTIONS:
Device: HR-pQCT — Xtreme CT® device is a high resolution peripheral quantitative computed tomography (HR-pQCT) used to measure bone density and quantify the bone architecture to 3D at the extremities of the human body.
  For the study, the device will be used to assess bone density and microarchitecture at the forearm and shin for a systemic effect. In rheumatoid arthritis, bone density and microarchitecture will also be measured at the metacarpophalangeal.
Device: DEXA — The Lunar Dual Energy X-ray Absorptiometry (DEXA) is a third generation multi-captor DEXA device that allow short duration measurements. It measures Bone Mineral Density (BMD) at the spine and the femoral neck
Device: pQCT — Peripheral Quantitative Computed Tomography (pQCT) will be performed and measure bone and muscle parameters.

SUMMARY:
Bone fracture occurrence is associated with an increasing of morbidity and mortality. Some factors of fracture occurrence have been highlighted. For example, some diseases or therapy are known to increased risk of bone fracture only in some patients. Accordingly, it is important for clinicians to identify patients at risk for bone fracture. Right now, various tools are available for the clinicians:

* clinical exam,
* bone mineral density assessed by Dual Energy X-ray Absorptiometry (DEXA),
* an algorithm based on interrogation, clinical exam and bone mineral density. However, prediction of bone fracture risk needs to be improved since only 50% of bone fractures can be predicted. DEXA provides information for fracture risk estimation, but it is unable to distinguish cortical part to trabecular part. It also fails to quantify the microstructural properties that influence bone strength. Bone microarchitecture, including the cortical compartment can now be assessed in vivo by the HR-pQCT. This technique allows access to several parameters: on the one hand the volumetric bone mineral density for the whole area measured as well as cortical and trabecular regions, and on the other hand, the thickness and cortical porosity and the number of trabecular, their orientation and distribution.

Thus, the HR-pQCT allows realizing a virtual bone biopsy and provides information on cortical and trabecular bone microarchitecture. This is the only noninvasive way to assess cortical and trabecular bone microarchitecture.

ELIGIBILITY:
Inclusion Criteria:

1. For patients:

   1.1.Women or Men taken in charge in Saint-Etienne' Hospital and one of the following pathologies: 1.1-a : Osteoporosis defined as: history of fracture by bone fragility documented 1.1-b : Bone Fragility: Patient with the indication of bone densitometry without a fracture history 1.1-c Articular inflammatory disease: Rheumatoid Arthritis, Spondyloarthritis 1.1-d Endocrine diseases : Primary Hyperparathyroidism, Constitutional Thinness, Anorexia nervosa 1.2. written consent
2. For controls:

2.1. Episode of acute back pain or radicular pain (lasting for less than a month) with taking corticosteroid less than 1 month 2.2. written consent

Exclusion Criteria:

drugs induced bone loss: 1.1.Anti-aromasine or GnRH agonist for at least 6 months, 1.2. Corticosteroid therapy 1.3. Antiepileptic carbamazepine, phenobarbital, phenytoin, primidone, valproic acid for at least 6 months) 2. fracture due to bone fragility 3. drug with bone effect (bisphosphonate, teriparatide, strontium ranelate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Bone microarchitecture parameter | Day 1
  Compare between patient group and control group bone microarchitecture parameter.
  Different bone microarchitecture parameter is a composite outcome assessed by HR-pQCT : Total volumetric mineral density (mg/ccm HA), Trabecular volumetric mineral density (mg/ccm HA), Cortical volumetric mineral density (mg/ccm HA), Trabecular number ((1/mm), Trabecular thickness (mm), Cortical thickness (mm), Trabecular separation (mm), Cortical porosity (%)

SECONDARY OUTCOMES:
Bone density | day 1
  Bone density is a composite outcome measured with three devices HR-pQCT, pQCT and DEXA.
  Parameters measured with HR-pQCT are : Total volumetric mineral density (mg/ccm HA), Trabecular volumetric mineral density (mg/ccm HA) and Cortical volumetric mineral density (mg/ccm HA).
  Parameters measured with pQCT are: total bone mineral content (mg), total bone surface (mm2), total bone density (mg/mm3), cortical and trabecular density (mg/mm3), and the bone resistance index (g2/mm).
  Parameter measured by DEXA is Bone Mineral Density (BMD, g/cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Thomas, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No